CLINICAL TRIAL: NCT05399901
Title: Use of Transabdominal M-mode Ultrasonography in the Assessment and Treatment of Pelviperineal Dysfunctions
Brief Title: M-mode Ultrasonography in the Assessment and Treatment of Pelviperineal Dysfunctions (PerineUM)
Acronym: PerineUM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, María Elena del Baño-Aledo, Principal Investigator, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PerineUM2022
Record Dates: First submitted 2022-05-23; First posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Pelvic Floor Disorders
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMG BFB (Experimental): An educational program will be implemented, and active exercises of the PFM will be performed using verbal instructions together with electromyographic biofeedback (BFB).
  Interventions: Other: Electromyographic biofeedback
- M-mode US (Experimental): An educational program will be implemented, and active exercises of the PFM will be performed using verbal instructions together with transabdominal M-mode ultrasound biofeedback (US).
  Interventions: Other: M-mode US biofeedback

INTERVENTIONS:
Other: Electromyographic biofeedback — Active exercises of the pelvic floor muscles and verbal instructions and EMG Biofeedback
  Arms: EMG BFB
Other: M-mode US biofeedback — Active exercises of the pelvic floor muscles and verbal instructions and M-mode Ultrasound Biofeedback
  Arms: M-mode US

SUMMARY:
Objectives: To analyze the Mode M ultrasound use in the assessment of pelvic floor musculature (PFM) and in the rehabilitation of motor control in pelviperineal dysfunctions that affect the support of pelvic organs, urinary and fecal continence and reproductive and sexual functions.

Methodology: A cross-sectional descriptive study will be followed by a randomized clinical trial. There will be two samples: a sample of volunteers without PFM dysfunction; and a sample of patients with pelviperineal dysfunction derived from health centers in the Region of Murcia. An intra- and interobserver reliability study of transabdominal M-mode ultrasound of PFM will be performed. Then, a cross-sectional descriptive study of the functional behavior of PFM will be used in different functional situations such as: voluntary contraction at maximum force, fast contraction, Valsalva maneuver and forced cough. The following ultrasound variables will be measured: direction and amount of displacement, speed of displacement and time of contraction. Correlations between ultrasound variables and sociodemographic and clinical variables will be analyzed. The randomized clinical trial will compare a PFM contraction awareness treatment based on endocavitary digital contact with a motor learning program based on transabdominal mode M ultrasound biofeedback.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pelvic floor dysfunction derived from the pelvic floor unit of HLA La Vega in the city of Murcia diagnosed by the doctor and without previous training in pelvic floor muscles contraction.

Exclusion Criteria:

* Pregnancy, a history of pelvic floor surgery in the previous year, neurological injury with affectation of the sacral reflex from S2 to S4, previous delivery in a period of less than 6 weeks or known or suspected urinary tract infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Changes in the self efficacy expectations in performing pelvic floor exercises. | At baseline and after the intervention (1 week from baseline)
  It will be assessed by the Broome Pelvic Muscle Self-Efficacy Scale (PMSES) Spanish version. Self-efficacy expectations, specifically for performing pelvic floor exercises, are measured with 14 items with responses between 0 and 100. One hundred represents high level of confidence.
Changes in the outcome expectations for pelvic-floor exercise treatment. | At baseline and after the intervention (1 week from baseline)
  It will be assessed by the Broome Pelvic Muscle Self-Efficacy Scale (PMSES) Spanish version. Outcome expectations are measured with 9 items with responses between 0 and 100. One hundred represents high level of confidence.

SECONDARY OUTCOMES:
Change in the displacement of the base of the bladder during voluntary contraction of the pelvic floor. | At baseline and after the intervention (1 hour from baseline)
  It will be measured by Ultrasonography.

CONTACTS AND LOCATIONS:
Overall Officials: MARIA ELENA DEL BAÑO ALEDO, PhD, Principal Investigator — Murcia University

IPD SHARING:
Plan to Share IPD: No